CLINICAL TRIAL: NCT02620137
Title: Maintenance of Multivitamin Supplements After Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HURJC15-15
Record Dates: First submitted 2015-11-26; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multicentrum® 3 months (Experimental): Patients maintaining the multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) during 3 months
  Interventions: Drug: Multicentrum® (Pfizer, Spain) 3 months
- Multicentrum® 12 months (Active Comparator): Patients maintaining the multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) during 12 months
  Interventions: Drug: Multicentrum® (Pfizer, Spain) 12 months

INTERVENTIONS:
Drug: Multicentrum® (Pfizer, Spain) 3 months — The multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) will be maintained during 3 months
  Other Names: Multicentrum 3 months
  Arms: Multicentrum® 3 months
Drug: Multicentrum® (Pfizer, Spain) 12 months — The multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) will be maintained during 12 months
  Other Names: Multicentrum 12 months
  Arms: Multicentrum® 12 months

SUMMARY:
A prospective randomized study of patients undergoing a laparoscopic sleeve gastrectomy was performed. Patients were randomized into 2 groups: those patients receiving the multivitamin supplement during 3 months (Group 1), and those receiving the supplement during 12 months (Group 2). Laboratory data were recorded: vitamins and oligoelements at 3, 6 and 12 months after surgery.

DETAILED DESCRIPTION:
A prospective randomized study of patients undergoing a laparoscopic sleeve gastrectomy was performed. Patients were randomized into 2 groups: those patients receiving the multivitamin supplement (Multicentrum, Pfizer, 1 tablet/day) during 3 months (Group 1), and those receiving the supplement during 12 months (Group 2). Laboratory data were recorded: vitamins (D, B12 and folic acid) and oligoelements (calcium, iron, phosphorus, magnesium and zinc) at 3, 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic sleeve gastrectomy
* BMI >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity

Exclusion Criteria:

* documented gastroesophageal reflux
* patients with uncontrolled psychiatric disorders
* active infections or malignancies
* any other concomitant pathology considered as a contraindication for bariatric surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Iron serum levels | 12 months
  Iron serum levels will be investigated in blood samples 12 months after surgery

SECONDARY OUTCOMES:
Calcium serum levels | 12 months
  Calcium serum levels will be investigated in blood samples 12 months after surgery
Vitamin B12 serum levels | 12 months
  Vitamin B12 serum levels will be investigated in blood samples 12 months after surgery
Folic acid serum levels | 12 months
  Vitamin B12 serum levels will be investigated in blood samples 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Duran, Study Director — Department of Surgery

REFERENCES:
- [Derived] Ruiz-Tovar J, Llavero C, Zubiaga L, Boix E; OBELCHE group. Maintenance of Multivitamin Supplements After Sleeve Gastrectomy. Obes Surg. 2016 Oct;26(10):2324-30. doi: 10.1007/s11695-016-2084-5. PMID 26843085